CLINICAL TRIAL: NCT04398576
Title: Primary Care Implementation Study to Scale up Early Identification and Brief Interventions and Reduce Alcohol Related Negative Outcomes at Community Level (PINO): Study Protocol for a Quasi-experimental 3-arm Study
Brief Title: Primary Care Implementation Study to Scale up EIBI and Reduce Alcohol Related Negative Outcomes
Acronym: PINO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Cathy Matheï, Professor, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: s63342
Record Dates: First submitted 2020-05-13; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Harmful; Use, Alcohol; Hazardous; Use, Alcohol
Keywords: Alcohol; Screening; Brief Intervention; Implementation; Training and Support; Primary Healthcare; Scaling up; Community actions; hazardous alcohol use heavy drinking; harmful use of alcohol; heavy drinking
MeSH Terms: interventions — Training Support; Community Participation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Support as usual (No Intervention): There will be no interventions, only support as usual. All GPs receive an information package by post or via e-mail containing:
  * Belgian guidelines on the management of hazardous and harmful alcohol use
  * A summary card about EIBI for hazardous and harmful alcohol consumption.
  * Internet links to documentation of the medical association and the Flemish centre of expertise on alcohol and drugs(31).
  An EHR-update allows the use of an extra e-form permitting standardised introduction of screening results from the Alcohol Use Disorders Identification Test (-Consumption) (AUDIT(-C)), alcohol-related diagnoses and actions including provision of oral brief advice/intervention, referral to a digital-based system for advice and/or referral to another health care provider.
- Training and support (Active Comparator): All GPs receive an information package by post or via e-mail containing:
  * Belgian guidelines on the management of hazardous and harmful alcohol use
  * A summary card about EIBI for hazardous and harmful alcohol consumption.
  * Internet links to documentation of the medical association and the Flemish centre of expertise on alcohol and drugs(31).
  An EHR-update allows the use of an extra e-form permitting standardised introduction of screening results from the Alcohol Use Disorders Identification Test (-Consumption) (AUDIT(-C)), alcohol-related diagnoses and actions including provision of oral brief advice/intervention, referral to a digital-based system for advice and/or referral to another health care provider.
  There shall be tailored training and support for the general practioners. At the start of the study, this group receives two face-to-face educational trainings of two hours each. Another two face-to-face booster sessions will follow at 6 and at 12 months.
  Interventions: Behavioral: Training and support
- Training and support and community actions (Active Comparator): In this group, GPs receive the same training and support as in the second arm (training and support). There will also be embedded community-based actions within a local strategy.
  Interventions: Behavioral: Training and support; Behavioral: Community actions

INTERVENTIONS:
Behavioral: Training and support — GP's receive the tools to make early identification of harmful and hazardous alcohol use possible. They are given guidelines to apply a brief intervention. At the start of the study, the T&S-group receives two face-to-face educational trainings of two hours each. Another two face-to-face booster sessions will follow at 6 and at 12 months.
  Arms: Training and support; Training and support and community actions
Behavioral: Community actions — There will be embedded community-based actions within a local strategy.
  Arms: Training and support and community actions

SUMMARY:
The aim of this implementation study is to compare the effect of tailored training and support (T&S) for general practioners with T&S and alcohol community actions and the impact it has on early identification of hazardous and harmful drinking and brief intervention.

DETAILED DESCRIPTION:
A quasi-experimental three-arm implementation study will be undertaken in Flanders (Belgium) to assess the effects of tailored training and support to general practitioners (GPs) alone or in an area context of alcohol community actions and compared to 'support as usual' on GP's performance in terms of early identification of hazardous and harmful drinking and brief intervention.

The study will last 18 months and will take place in three cities of comparable size. In each area at least 28 GPs will be recruited.

The primary outcome will be the proportion of consulting adult patients screened for hazardous and harmful alcohol use at the end-point of an 18-month implementation period. The secondary outcomes will be the screening rate as assessed at 3, 6, 9, 12 and 15 months and the proportion of patients screening positive for hazardous and harmful alcohol use that receive a brief intervention at 3,6,9, 12, 15 and 18 months. Furthermore, the relation between GP's views and needs and practices' contexts, and EIBI performance will be explored.

Data regarding screening and brief intervention activities will be collected from the electronic health records (EHR).

ELIGIBILITY:
Inclusion Criteria:

* GP or GP trainee
* Dutch language use in practice
* Working in general practice in 3 cities of comparable size or their sub municipalities

Exclusion Criteria:

- No possibility of integration of e-form into the EHR-system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Early Identification Rate (EIR) | 18 months
  The Primary outcome or the Early Identification Rate (EIR) is the proportion of adult consulting patients (18 years and over) that is screened for alcohol consumption during a period of 18 months per area.

SECONDARY OUTCOMES:
EIR every 3 months | at 3, 6, 9, 12 and 15 months
  The Early Identification Rate (EIR) assessed at 3, 6, 9, 12 and 15 months per area.
BIR | at 3, 6, 9, 12, 15 and 18 months
  The Brief Intervention rate (BIR) is the proportion of patients screening positive for hazardous or harmful alcohol use that received oral brief advice/intervention and/or were referred to digital-based system for advice, and/or were referred to another provider assessed at 3, 6, 9, 12, 15 and 18 months per area.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Matheï, master, Principal Investigator — professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pussig B, Pas L, Li A, Vermandere M, Aertgeerts B, Mathei C. Primary care implementation study to scale up early identification and brief intervention and reduce alcohol-related negative outcomes at the community level (PINO): study protocol for a quasi-experimental 3-arm study. BMC Fam Pract. 2021 Jul 1;22(1):144. doi: 10.1186/s12875-021-01479-9. PMID 34210261